CLINICAL TRIAL: NCT02265627
Title: Pharmacokinetics, Safety and Tolerability of Single Dose BIIL 284 BS in Patients With Hepatic Impairment in Comparison to Healthy Subjects (An Open Label, Matched Pair, Two Center Study)
Brief Title: Pharmacokinetics, Safety and Tolerability of BIIL 284 BS in Patients With Hepatic Impairment in Comparison to Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 543.26
Record Dates: First submitted 2014-10-15; First posted 2014-10-16 (Estimated); Last update posted 2014-10-16 (Estimated); Status verified 2014-10

CONDITIONS: Hepatic Insufficiency
MeSH Terms: conditions — Hepatic Insufficiency | interventions — amelubant

ARMS (3):
- BIIL 284 BS, normal hepatic function (Experimental)
  Interventions: Drug: BIIL 284 BS
- BIIL 284 BS, mild hepatic impairment (Experimental)
  Interventions: Drug: BIIL 284 BS
- BIIL 284 BS, moderate hepatic impairment (Experimental)
  Interventions: Drug: BIIL 284 BS

INTERVENTIONS:
Drug: BIIL 284 BS

SUMMARY:
To investigate the pharmacokinetics of a single dose of BIIL 284 BS in patients with hepatic impairment in comparison to healthy subjects

ELIGIBILITY:
Inclusion Criteria:

Healthy Subjects

* Written informed consent signed and dated prior to participation into the study (including medication washout)
* Male of female 24-70 years of age
* All subjects should be within (+- 20 %) of their ideal body weight (Broca-Index)
* Healthy subjects must be able to be comparably matched to a hepatic impaired patient according to age (+- 5 years), weight (+- 30 lbs), gender, and smoking status
* Volunteers will have no evidence of clinically relevant concomitant disease based upon the following: a detailed medical and surgical history, a complete physical examination including vital signs, 12-lead ECG, complete blood count (CBC) with differential and platelets, prothrombin time (PT), blood chemistry, hematology and urinalysis
* Female subjects need to be of non-childbearing potential (post-menopausal), tubal ligation or total hysterectomy) and had to provide a negative pregnancy test at the screening visit or subjects is a male
* Tested negative at the screening visit for the following drug screen panel (barbiturates, benzodiazepines, amphetamines, opiates, cocaine, cannabinoids)

Patients with hepatic impairment

* Written informed consent signed and dated prior to participation into the study (including medication washout)
* Male of female 24-70 years of age
* All subjects should be within (+- 20 %) of their ideal body weight (Broca-Index)
* Proven history of cirrhosis confirmed by liver/spleen scan or biopsy (within one year)
* Hepatic impairment: A Child-Pugh classification of Class A, or B
* Volunteers will have no evidence of clinically relevant concomitant disease (other than hepatic impairment) based upon the following: a detailed medical and surgical history, a complete physical examination including vital signs, 12-lead ECG, CBC with differential and platelets, prothrombin time (PT), blood chemistry, hematology and urinalysis
* Tested negative at the screening visit for the following drug screen panel (barbiturates, benzodiazepines, amphetamines, opiates, cocaine, cannabinoids). Unless known drugs were being used for medicinal reasons. For this reason the sponsor and investigator were notified
* Female patients were of non-childbearing potential (post-menopausal), tubal ligation or total hysterectomy) and had to provide a negative pregnancy test at the screening visit

Exclusion Criteria:

Healthy subjects

* Tested positive for Hepatitis B surface antigen, Hepatitis C antibody or HIV antibody
* Have a significant acute or chronic disease, which could have interfered with the objectives of the study
* Small or difficult to locate arm or hand veins that would impair the clinician's ability to draw multiple blood samples or to place a venous catheter
* Likely to need concomitant medication during the study period, which could interfere with the objectives of the study
* Had given a blood donation during the month preceding the study drug administration
* Alcohol consumption > 2 drinks daily (one drink defined as: 12 ounces of beer, 4 ounces of wine or 1.5 ounces of spirits)
* Coffee or tea consumption > 3 cups per day or xanthine containing drinks > 0.5 liter/day
* History of any clinically significant hematological, respiratory, cardiovascular, renal or central nervous system (CNS) disease or other medical condition that is capable of altering the metabolism or elimination of drugs, or of constituting a risk factor when taking the study drug
* History of drug addiction or alcoholism
* Any medical or psychological condition which could relapse during or immediately after the study
* Use of any drug or nutrient which could induce or inhibit hepatic microsomal enzymes within one month of the start of the study or longer based on the elimination half-life of the drug
* Use of experimental new drug one month prior to study drug administration
* Consumed any medicine whatsoever (including over the counter (OTC) drugs) within two weeks of the scheduled administration of the study drug

Patients with Hepatic Impairment

* Positive serology for HIV
* Have a significant acute or chronic disease (except hepatic disease), which is unstable or could interfere with the objectives of the study
* Small or difficult to locate arm or hand veins that would impair the clinician's ability to draw multiple blood samples or to place a venous catheter
* Have hepatocellular carcinoma, extrahepatic biliary obstruction, surgical portal-systemic shunting, acute hepatitis of any origin
* Digestive bleeding within one month of inclusion
* Likely to need concomitant medication during the study period, which could interfere with the objectives of the study
* Had given a blood donation during the month preceding study entry
* Coffee or tea consumption > 3 cups per day or xanthine containing drinks > 0.5 liter/day
* History of any clinically significant hematological, respiratory, cardiovascular, renal or CNS disease or other medical condition (except hepatic impairment) that is capable of altering the metabolism or elimination of drugs, or of constituting a risk factor when taking the study drug
* Any medical or psychological condition which could relapse during or immediately after the study
* Use of any drug or nutrient which could induce or inhibit hepatic microsomal enzymes within one month of the start of the study or longer based on the elimination half-life of the drug
* Use of experimental new drug within the previous month

Ages: 24 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2000-03; Primary Completion 2000-09 (Actual)

PRIMARY OUTCOMES:
Plasma concentration-time profiles of the analytes at different time points | Up to 84 hours after drug administration

SECONDARY OUTCOMES:
Maximum measured concentration of BIIL 315 ZW in plasma (Cmax) | Up to 84 hours after drug administration
Time from dosing to the maximum concentration of BIIL 315 ZW in plasma (tmax) | Up to 84 hours after drug administration
Area under the concentration-time curve of BIIL 315 ZW in plasma at different time points (AUC) | Up to 84 hours after drug administration
Terminal half-life of BIIL 315 ZW in plasma (t1/2) | Up to 84 hours after drug administration
Total mean residence time of BIIL 315 ZW in the body (MRTtot) | Up to 84 hours after drug administration
Total apparent clearance of BIIL 315 ZW in plasma after oral administration (CLtot/F) | Up to 84 hours after drug administration
Apparent volume of distribution during the terminal phase λz following an extravascular dose (Vz/F) | Up to 84 hours after drug administration
Number of patients with clinically relevant findings in vital signs | Up to 4 days after drug administration
  blood pressure, pulse rate
Changes from baseline in spirometry | Pre-dose and 1 hour after drug administration
Number of patients with clinically relevant findings in laboratory tests | Up to 4 days after drug administration
Number of patients with clinically relevant findings in 12-lead ECG | Up to 4 days after drug administration
Changes from baseline in physical examination | Pre-dose and 4 days after drug administration
Number of patients with adverse events | Up to 11 days after drug administration